CLINICAL TRIAL: NCT01765036
Title: Contrast-harmonic Endoscopic Ultrasound (CH-EUS) for the Diagnosis of Pancreatic Adenocarcinoma: Results of the First Multicenter Prospective Study With Intra- and Interobserver Concordances Evaluation
Brief Title: Contrast-harmonic Endoscopic Ultrasound (CH-EUS) for the Diagnosis of Pancreatic Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, Gincul Rodica, MD, Société Française d'Endoscopie Digestive
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-004676-44
Record Dates: First submitted 2013-01-03; First posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: contrast-enhanced endoscopic ultrasound; pancreatic adenocarcinoma
MeSH Terms: interventions — contrast agent BR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SonoVue® (Experimental): Non randomised study
  Sonovue 4,8 ml intravenous administration, in 1 bolus, during the EUS examination
  Interventions: Drug: SonoVue®

INTERVENTIONS:
Drug: SonoVue® — An intravenous 4.8 ml SonoVue® bolus injection was administered to each patient during the procedure
  Other Names: soufre hexafluorure

SUMMARY:
Ductal adenocarcinoma is the most frequent pancreatic solid lesion and the most common tumor of the pancreas. Given its poor prognosis and the major therapeutic consequences, the discrimination between PA and other pancreatic solid lesions is mandatory. EUS is admitted as the most sensitive imaging procedure for the detection and characterization of pancreatic tumors [1-3]. Nevertheless it remains difficult to differentiate, on morphological features, PA from other solid masses. For 15 years, endoscopic ultrasound fine needle aspiration (EUS-FNA) has demonstrated its efficiency for tissue sampling and cyto-histologic diagnosis of PA. However, the negative predictive value (NPV) for the diagnosis of pancreatic adenocarcinoma (PA) remains low (30-70%) in the published prospective series [4]. So, in case of negative result, the choice between surgery and follow-up remains difficult. Additional criteria to get the decision are then warranted.

The assessment of pancreatic tumor enhancement using ultrasound contrast agents (UCAs) in real time with imaging specific methods seems useful to improve their characterization [4-8] either by contrast-enhanced EUS (CE-EUS) or, more recently, by contrast-enhanced harmonic EUS (CH-EUS).

The aims of this prospective multicenter study is:

1. to compare the NPV of contrast-enhanced endoscopic ultrasound (CH-EUS) and EUS-FNA for the diagnosis of PA;
2. to assess the intra- and inter-observer concordances of CH-EUS for the diagnosis of PA.

DETAILED DESCRIPTION:
100 patients with a solid pancreatic mass of indeterminate origin must be prospectively included in 3 French centers Exclusion criteria: presence of a cystic component greater than 25 % of the total volume of the lesion, pregnancy, lactation, age <18 years, and usual contraindications to SonoVue® injection.

All EUS procedure will be performed by 5 experienced endosonographers as follows:

1. Conventional gray-scale B-mode and conventional power Doppler EUS to assess the EUS characteristics of the pancreatic lesion (localization, size, echogenicity, cystic component), the aspect of the surrounding parenchyma as well as the presence of proximal duct dilation, vessels infiltration, and collateral veins; tumor and nodes (uTN) staging. A systematic video of the 2 modes will be recorded.
2. CH-EUS will be performed to assess the microvascularization of the lesion and of the surrounding parenchyma: the echoendoscope will be placed in front of the pancreatic lesion and the contrast-specific mode will be engaged with simultaneous monitoring by fundamental B mode. A mecanical index (MI) of 0.4 will be chose based on previous studies [4-6]. An intravenous 4.8 ml SonoVue® bolus injection will be administrated through an antecubital vein, using a 20 Gauges catheter, followed by 20 ml saline flush. Examination of pancreatic lesion will be evaluated in real time and a video of each examination will be record and store. The examination lasted up to 3 minutes after SonoVue® injection to ensure full examination of the lesion in arterial (hyper echogenicity of the aorta, superior mesenteric, hepatic or splenic arteries) and venous phases (hyper echogenicity of the splenic-mesenteric-portal vessels). The pancreatic lesion enhancement pattern will be compare to the adjacent pancreatic parenchyma. We differentiated 3 patterns: hypo-, iso- or hyperenhancement. The operator classified the lesion as pancreatic adenocarcinoma (PA) or non PA. Based on previous pilot studies, lesion in hypoenhancement consider as PA while lesion in hyper or isoenhancement as non-PA [4-6]. In case of tumors with mixed pattern the lesion was considered as PA if a significant area (>10% of the surface) is in hypoenhancement.
3. EUS-FNA: a specimen will be obtain from all lesions using a 22 Gauge needle. Final diagnosis will be based on pathological findings obtained either surgically or by EUS-FNA. In the absence of histological evidence, follow-up (F-U) of patients for 12 months will be carried out. The diagnosis of PA ruled out if no sign of malignancy (disease regression or absence of disease progression) present at the end of F-U.
4. Images reviewing: at the end of the study an anonymous digital video recording of each procedure including B mode, power Doppler mode and CHE mode will be performed.

Statistical analysis. The McNemar test will be use to compare the CH-EUS performance for the diagnosis of PA to EUS-FNA and final diagnosis. Sensitivity (Se), specificity (Spe), predictive positive value (PPV), negative predictive value (NPV) and accuracy with 95% confidence intervals (95%CI) will be calculate. A p value of 0.05 considered statistically significant. Intra- and interobserver agreements of CH-EUS for the diagnosis of PA will assess using kappa statistics and associated 95% CI. Depending on Kappa values, agreement will considered as minor (0.01-0.20), fair (0.21-0.40), moderate (0.41-0.60), high (0.61-0.80), or almost perfect (0.81-1.00), beyond chance.

ELIGIBILITY:
Inclusion Criteria:

* patients with a solid pancreatic mass of indeterminate origin

Exclusion Criteria:

* presence of a cystic component greater than 25 % of the total volume of the lesion, pregnancy, lactation, age <18 years, and usual contraindications to SonoVue® injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
negative predictive value (NPV) of contrast-enhanced endoscopic ultrasound (CH-EUS) for the diagnosis of pancreatic adenocarcinoma (PA) | one year
  To evaluate the NPV of CH-EUS for the diagnosis of PA to EUS-FNA and final diagnosis

SECONDARY OUTCOMES:
to asses intra-observer concordances of CH-EUS for the diagnosis of PA | two days
  an anonymous digital video recording of each procedure including B mode, power Doppler mode and CHE mode was created. A 2-days joint work session was organized with 7 endosonographers: the 5 senior endoscopists who had performed the examinations and 2 juniors. To harmonizing the interpretation a short teaching session was done with some cases not included in the series. The different types of enhancement of solid pancreatic masses histologically proven (PA, benign and malignant NET, pancreatic metastases, and focal mass of CP) were shown. During day 1 the 7 operators reviewed independently and in a random order all 100 anonymous videotapes. One senior and 1 junior reviewed all videotapes a second time in a different random order. Each observer had to independently classify the lesion as PA or not. During day 2 a joint review was done with the cases where a discrepancy of interpretation has been observed. A final consensus for the diagnosis was proposed if possible.
to asses inter-observer concordances of CH-EUS for the diagnosis of PA | two days
  an anonymous digital video recording of each procedure including B mode, power Doppler mode and CHE mode was created. A 2-days joint work session was organized with 7 endosonographers: the 5 senior endoscopists who had performed the examinations and 2 juniors. To harmonizing the interpretation a short teaching session was done with some cases not included in the series. The different types of enhancement of solid pancreatic masses histologically proven (PA, benign and malignant NET, pancreatic metastases, and focal mass of CP) were shown. During day 1 the 7 operators reviewed independently and in a random order all 100 anonymous videotapes. One senior and 1 junior reviewed all videotapes a second time in a different random order. Each observer had to independently classify the lesion as PA or not. During day 2 a joint review was done with the cases where a discrepancy of interpretation has been observed. A final consensus for the diagnosis was proposed if possible.
sensibility (Se) of contrast-enhanced endoscopic ultrasound (CH-EUS) for the diagnosis of pancreatic adenocarcinoma (PA) | one year
  To evaluate the Se of CH-EUS for the diagnosis of of pancreatic adenocarcinoma (PA) to EUS-FNA and final diagnosis
Specificity (Spe) of CH-EUS for the diagnosis of pancreatic adenocarcinoma (PA) | one year
  To evaluate the specificity (Spe) of CH-EUS for the diagnosis of PA to EUS-FNA and final diagnosis
Positive predictive value (PPV) of CH-EUS for diagnosis of pancreatic adenocarcinoma (PA) | one year
  To evaluate the PPV of CH-EUS for the diagnosis of PA to EUS-FNA and final diagnosis
Accuracy of CH-EUS for the diagnosis of PA | one year
  To evaluate the accuracy of CH-EUS for the diagnosis of PA to EUS-FNA and final diagnosis value (PPV)
Accuracy of CH-EUS compared to EUS-FNA | one year
  To compare the accuracy of CH-EUS and EUS-FNA for the diagnosis of PA with 95% confidence intervals (95%CI)

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Gincul, MD, Principal Investigator — Société Française d'Endoscopie Digestive; Bertrand Napoleon, MD, Study Chair — Société Française d'Endoscopie Digestive
Locations (1):
- Société Française d'Endoscopie Digrestive, Paris, France